CLINICAL TRIAL: NCT05617651
Title: Phase 1 Study to Evaluate the Safety and the Pharmacokinetics of IY-NT-T in Healthy Adult Volunteers Under Fed Condition
Brief Title: Study to Evaluate the Safety and the Pharmacokinetics of IY-NT-T
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Il-Yang Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DTC22-IP018
Record Dates: First submitted 2022-11-08; First posted 2022-11-15 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Pharmacokinetics
Keywords: proton pump inhibitor

STUDY DESIGN:
Masking Description: In order to prevent distortion (bias) affecting test results during sample analysis, this clinical trial shall not be disclosed to analysis manager and analyst until the specimen analysis is completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A group (Active Comparator): Period 1 : Ilaprazole 10mg 2Tab, one a day
  Period 2 : Ilaprazole 20mg 1Tab, one a day
  Period 3 : Ilaprazole 10mg 2Tab, one a day
  Interventions: Drug: IY-NT-T; Drug: IY-NT-R
- B group (Active Comparator): Period 1 : Ilaprazole 20mg 1Tab, one a day
  Period 2 : Ilaprazole 10mg 2Tab, one a day
  Period 3 : Ilaprazole 20mg 1Tab, one a day
  Interventions: Drug: IY-NT-T; Drug: IY-NT-R

INTERVENTIONS:
Drug: IY-NT-T — Ilaprazole 20mg
Drug: IY-NT-R — Ilaprazole 10mg
  Other Names: Noltec(the brand name)

SUMMARY:
This study evaluate the pharmacokinetic and safety of IY-NT-T in healthy adults

DETAILED DESCRIPTION:
Phase 1 study to evaluate the safety and the pharmacokinetics of IY-NT-T in healthy adult volunteers under fed condition

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers aged 19 years and above at screening
2. A volunteer who weighs ≥ 50kg (≥ 45kg for women) and has a body mass index(BMI)* of ≥18.0 and ≤ 30 at screening

   *BMI(body mass index, kg/m^2)= Body weight (kg)/[height (m)^2]
3. A volunteer who has no congenital or chronic diseases, no pathological symptoms, or findings from medical examination at screening
4. A volunteer who is determined by the principal investigator or sub-investigator(responsible physician) as eligible as a subject based on diagnostic tests( hematology, hematochemical, serum, urinalysis) and electrocardiogram tests established and conducted according to the characteristics of the study drug
5. A volunteer and their spouse or partner, who agree to use a medically appropriate method of contraception to exclude potential of pregnancy and not to provide sperm or ova from the first dose to 7 days after the last dose of study drug

   * Contraception methods: Intrauterine device, vasectomy, tubal ligation and contraceptive barrier methods (male condoms, women condoms, cervical caps. Contraceptive diaphragm, sponge,etc) used in combination or if spermicide is used, two or more contraceptive barrier methods
6. A volunteer who voluntarily provided written consent to participation in the entire study process after being fully informed of the study objective, contents, characteristics of the study drugs, and expected adverse reactions, prior to study participation

Exclusion Criteria:

1. A volunteer who has a history or present symptoms of clinically significant disorders relating to any of the following: digestive system, cardiovascular system, endocrine system, respiratory system, blood and lymphatic, infectious disease, renal, urinary, and reproductive, system, nervous system, musculoskeletal system, immune system, otolaryngology, skin and subcutaneous tissue system, and ophthalmic system
2. A volunteer who has a history of gastrointestinal surgery that may affect drug absorption (except simple appendectomy or hernia surgery) or has gastrointestinal diseases
3. A volunteer who has taken drugs that induce or inhibit drug metabolizing enzymes such as barbiturates within 1 month prior to the first dose or who has taken drugs that may interfere with clinical study within 10 days prior to the first dose(Provided that, participation may be considered based on drug-drug interaction, pharmacokinetics and pharmacodynamics(such as half-life) of study drug)
4. A volunteer who has participated in other clinical trials or bioequivalence studies within 6 months prior to the first dose of the study drug
5. A volunteer who has participated in whole blood donation within 8 weeks prior to first dose, or apheresis donation within w weeks prior to first dose, or received blood donation within 4 weeks prior to first dose.
6. A volunteer that meets any of the following conditions within 1 month prior to first dose

   * Average alcohol intake(for men): > 21 glass/week
   * Average alcohol intake(for women): > 14 glass/week (1 glass = 50ml of soju or 30ml of liquor, or 250ml of beer)
   * Average cigarette smoking: > 20 cigarettes per day.
7. A volunteer that meets any of the following categories

   * Volunteer who is hypersensitive to the active ingredient or other ingredients of this drug
8. Patients that meet any of the following conditions

   * Gastric ulcer patients possibly related to a malignant tumor
   * Hepatic disorder or renal disorder patients
   * Patients receiving Atazanavir
   * Patients receiving Rilpivirine-containing products
9. A volunteer who is considered by the investigator to be ineligible to participate in this study for other reasons
10. Pregnant or nursing women

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2024-12-10 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Ilaprazole AUCt | Predose(0hour), after dose 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25, 26, 27, 28, 29, 30, 32, 34, 36, 40, 48 hour
  ilaprazole AUCt(Area under the concentration-time curve)
Ilaprazole Cmax | Predose(0hour), after dose 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25, 26, 27, 28, 29, 30, 32, 34, 36, 40, 48 hour
  ilaprazole Cmax(Maximum concentration of drug in plasma)

SECONDARY OUTCOMES:
Ilaprazole AUC∞ | Predose(0hour), after dose 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25, 26, 27, 28, 29, 30, 32, 34, 36, 40, 48 hour
  ilaprazole AUC∞(Area under the plasma drug concentration-time curve from time 0 to infinity)
Ilaprazole tmax | Predose(0hour), after dose 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25, 26, 27, 28, 29, 30, 32, 34, 36, 40, 48 hour
  ilaprazole tmax(Time to maximum plasma concentration)
Ilaprazole t1/2 | Predose(0hour), after dose 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25, 26, 27, 28, 29, 30, 32, 34, 36, 40, 48 hour
  ilaprazole t1/2(Terminal elimination half-life)
Ilaprazole tmax-tlag | Predose(0hour), after dose 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25, 26, 27, 28, 29, 30, 32, 34, 36, 40, 48 hour
  Ilaprazole tmax-tlag (Time to maximum plasma concentration minus Lag time)
Ilaprazole intra-subject tlag difference | Predose(0hour), after dose 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25, 26, 27, 28, 29, 30, 32, 34, 36, 40, 48 hour
  Ilaprazole intra-subject Lag time difference

CONTACTS AND LOCATIONS:
Overall Officials: Jae Woo Kim, MD, PhD, Principal Investigator — H Plus Yangji Hospital
Locations (1):
- H plus Yangji Hospital, Seoul, Gwanak-gu, South Korea

IPD SHARING:
Plan to Share IPD: No